CLINICAL TRIAL: NCT00151801
Title: Safety and Tolerability of Oral Two-Doses Estroprogestins Associated With Interferon-Beta 1a in Patients With Relapsing-Remitting Multiple Sclerosis
Brief Title: Safety and Tolerability of Interferon-Beta-1a and Estroprogestins Association in MS Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: S. Andrea Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NEU - PIL - 03
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2005-09-09 (Estimated); Status verified 2005-09

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; estroprogestins; interferon-beta; sex hormones; MRI
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1a

INTERVENTIONS:
Drug: estroprogestins
Drug: interferon-beta 1a

SUMMARY:
Clinical and experimental evidences suggests an immunomodulatory effect of sex hormones in multiple sclerosis.

The role of oral estroprogestins in the pathogenesis and in the clinical course of the disease is actually unknown.

The aim of the study is to investigate safety and tolerability of association of estroprogestins in two different doses with interferon-beta 1a in patients with relapsing-remitting multiple sclerosis.

DETAILED DESCRIPTION:
Phase 2, randomised, single blind, three arms study.

Follow-up of 24 months.

The study will include relapsing-remitting multiple sclerosis female patients.

Patients will be equally randomised into three groups: 1) patients treated with IFN-beta 1a (44 mcg for three times a week), 2) patients treated with IFN-beta 1a and lower-dose estroprogestins (desogestrel 150 mcg, etinilestradiol 20 mcg), 3) patients treated with IFN-beta 1a and higher-dose estroprogestins (desogestrel 25 mcg, etinilestradiol 40 mcg).

Safety and tolerability of the treatment will be evaluated using neurological examination and MRI analysis.

A complete neurological examination (with EDSS) will be performed at month 0, 6, 12, 18 and 24.

MRI examination will be assessed at baseline and at month 12 and 24. In the same day of MRI examination we'll collect blood samples for hormonal analysis (we'll measure sex hormones in the follicular and in the luteal phase of a single menstrual cycle).

During the follow-up patients will be evaluated also with: MS-Functional Composite at month 0, 6, 12, 18, 24; neuropsychological evaluation at month 0, 12, 24; Fatigue Severity Scale at month 0, 12, 24; Hamilton Depression Scale at month 0, 12, 24; Quality of Life scale (MSQOL54) at month 0, 12, 24.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* Clinically definite relapsing-remitting MS according to the McDonald criteria
* Age between 18-40 y.o.
* EDSS from 0 to 4.0, inclusive

Exclusion Criteria:

* History of migraine or thromboembolic events
* Reproductive system disorders
* Pregnancy or suspension of pregnancy within 12 months prior to randomisation
* Prior use of estroprogestins within the last 3 months prior to randomisation
* Prior use of immunosuppressive drugs within the last 12 months prior to randomisation
* Prior use of immunomodulating drugs within the last 6 months prior to randomisation
* Prior use of corticosteroids within the last 3 months prior to randomisation
* Have clinical relapse 30 days prior to randomisation

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200
Dates: Start 2002-05; Study Completion 2008-12

PRIMARY OUTCOMES:
Safety assessment at 6, 12, 18 and 24 months, including adverse events, physical examination and laboratory parameters
Relapse rate at 6, 12, 18 and 24 months,
EDSS progression at 12 and 24 months,
MS functional composite score at 12 and 24 months,

SECONDARY OUTCOMES:
Number and volume of new gad-enhancing lesions at 12 and 24 months
Number of new T1 and T2 lesions at 12 and 24 months
Brain volume changes at 12 and 24 months
Neuropsychological examination at 0, 12, 24 months
Hamilton scale for depression score at 0, 12, 24 months
MS Quality of Life scale score(MSQOL54)at 0, 12, 24 months
Fatigue Severity Scale score at 0, 12, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Tomassini, MD, Study Chair — Department of Neurological Science University of Rome "La Sapienza"; Fabiana Marinelli, MD, Principal Investigator — Department of Neurological Science, University of Rome "La Sapienza"; Carlo Pozzilli, MD, Study Director — Department of Neurological Science, University of Rome "La Sapienza"
Locations (1):
- Department of Neurology - University of Rome La Sapienza, Rome, Rome, Italy

REFERENCES:
- [Background] Hawkins SA, McDonnell GV. Benign multiple sclerosis? Clinical course, long term follow up, and assessment of prognostic factors. J Neurol Neurosurg Psychiatry. 1999 Aug;67(2):148-52. doi: 10.1136/jnnp.67.2.148. PMID 10406979
- [Background] Zorgdrager A, De Keyser J. Menstrually related worsening of symptoms in multiple sclerosis. J Neurol Sci. 1997 Jul;149(1):95-7. doi: 10.1016/s0022-510x(97)05396-3. PMID 9168172
- [Background] Bansil S, Lee HJ, Jindal S, Holtz CR, Cook SD. Correlation between sex hormones and magnetic resonance imaging lesions in multiple sclerosis. Acta Neurol Scand. 1999 Feb;99(2):91-4. doi: 10.1111/j.1600-0404.1999.tb00663.x. PMID 10071166
- [Background] Kim S, Liva SM, Dalal MA, Verity MA, Voskuhl RR. Estriol ameliorates autoimmune demyelinating disease: implications for multiple sclerosis. Neurology. 1999 Apr 12;52(6):1230-8. doi: 10.1212/wnl.52.6.1230. PMID 10214749
- [Background] Hernan MA, Hohol MJ, Olek MJ, Spiegelman D, Ascherio A. Oral contraceptives and the incidence of multiple sclerosis. Neurology. 2000 Sep 26;55(6):848-54. doi: 10.1212/wnl.55.6.848. PMID 10994007
- [Background] Randomised double-blind placebo-controlled study of interferon beta-1a in relapsing/remitting multiple sclerosis. PRISMS (Prevention of Relapses and Disability by Interferon beta-1a Subcutaneously in Multiple Sclerosis) Study Group. Lancet. 1998 Nov 7;352(9139):1498-504. PMID 9820297
- [Background] De Cicco Nardone F, Rossiello F, Iacopino F, Benedetto MT, Cinque B, Dell'Acqua S, Sica G. Effects of interferon-beta on steroid receptors, prostaglandins and enzymatic activities in human endometrial cancer. Anticancer Res. 1996 Jan-Feb;16(1):161-9. PMID 8615603
- [Background] Pozzilli C, Tomassini V, Marinelli F, Paolillo A, Gasperini C, Bastianello S. 'Gender gap' in multiple sclerosis: magnetic resonance imaging evidence. Eur J Neurol. 2003 Jan;10(1):95-7. doi: 10.1046/j.1468-1331.2003.00519.x. PMID 12535003
- [Derived] De Giglio L, Marinelli F, Barletta VT, Pagano VA, De Angelis F, Fanelli F, Petsas N, Pantano P, Tomassini V, Pozzilli C. Effect on Cognition of Estroprogestins Combined with Interferon Beta in Multiple Sclerosis: Analysis of Secondary Outcomes from a Randomised Controlled Trial. CNS Drugs. 2017 Feb;31(2):161-168. doi: 10.1007/s40263-016-0401-0. PMID 27995531